CLINICAL TRIAL: NCT02435251
Title: Changes in Anthropometry Following Ambulatory Orthopaedic Surgery
Acronym: CAS
Status: Withdrawn | Type: Observational
Why Stopped: study was no longer feasible
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leslie Bisson, June A. & Eugene R. Mindell, MD Professor and Chair, State University of New York at Buffalo
Other Study IDs: 458943-7
Record Dates: First submitted 2015-04-27; First posted 2015-05-06 (Estimated); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Knee Surgery; Shoulder Surgery
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: dual energy X-ray absorptiometry

SUMMARY:
The purpose of this research is to study changes in weight, body mass index, and percentage of fat following orthopaedic knee or shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years-old
* scheduled to undergo knee or shoulder ambulatory surgery

Exclusion Criteria:

* weighs greater than 350 pounds
* pregnancy
* history of bariatric surgery
* dieting or engaged in a weight loss program
* taking weight loss supplements
* undergoing other types of surgery during study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to undergo ambulatory orthopaedic surgery at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Fat mass | 6-weeks after surgery

SECONDARY OUTCOMES:
Lean mass | 6-weeks after surgery
Weight | 6-weeks after surgery
Body mass index | 6-weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Bisson, MD, Principal Investigator — University at Buffalo
Locations (1):
- UBMD Orthopaedics & Sports Medicine, Amherst, New York, United States